CLINICAL TRIAL: NCT01934010
Title: AM-101 in the Post-Acute Treatment of Peripheral Tinnitus 1 (AMPACT1) - an Open-Label Extension to the TACTT2 Study
Brief Title: AM-101 in the Treatment of Post-Acute Tinnitus 1
Acronym: AMPACT1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Auris Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AM-101-CL-12-03
Record Dates: First submitted 2013-08-15; First posted 2013-09-04 (Estimated); Results first posted 2018-03-09 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-04

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — PDCD5 protein, rat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AM-101 injection (Experimental): AM-101 gel for intratympanic injection
  Interventions: Drug: AM-101

INTERVENTIONS:
Drug: AM-101 — AM-101 gel for intratympanic injection

SUMMARY:
The purpose of this research study is to test the safety and local tolerance of repeated treatment cycles of AM-101.

DETAILED DESCRIPTION:
This open-label extension study is assessing the safety and local tolerance of repeated treatment cycles of AM-101 in subjects previously treated in the scope of the TACTT2 study (NCT01803646).

ELIGIBILITY:
Inclusion Criteria:

* Completion of TACTT2 study;
* Negative pregnancy test (woman of childbearing potential);
* Willing and able to attend the study visits during at least one treatment cycle.

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Adverse event leading to treatment discontinuation in TACTT2;
* Meniere's Disease, endolymphatic hydrops, acoustic neuroma, severe or fluctuating hearing loss, otitis media, otitis externa, abnormality of tympanic membrane;
* Ongoing drug-based therapy for otitis media or otitis externa;
* Drug-based therapy known as potentially tinnitus-inducing;
* Other treatment of tinnitus;
* Drug abuse or alcoholism;
* Subjects with psychiatric diseases requiring drug treatment;
* Use of antidepressant or anti-anxiety medication;
* Any clinically relevant disorder or abnormality in physical examination;
* Women who are breast-feeding, pregnant or who are planning to become pregnant during the study;
* Women of childbearing potential who are unwilling or unable to practice contraception.

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2014-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 260 subjects were enrolled and 257 subjects were treated in overall 59 active sites in Canada (6), the United States (35), the Czech Republic (7), Israel (2), Turkey (3) and Republic of South Korea (6). Subjects could only participate if they had been previously enrolled and completed the participation in the TACTT2 study.
Pre-assignment Details: Main Inclusion Criteria:
  * completion of TACTT2 study
  * negative pregnancy test (women of childbearing potential)
  * willing and able to attend the study visits during at least one treatment cycle.
Groups:
- 1 Cycle AM-101: Subjects participated in 1 treatment cycle and received one round of 3 repeated doses of AM-101 gel (0.87 mg/mL) within 5 days (D0-D4)
- 2 Cycles AM-101: Subjects that participated in 2 treatment cycles of the AMPACT1 study, received 3 repeated doses of AM-101 gel (0.87 mg/mL) within 5 days (D0 - D4) in cycle 1 and after final follow-up (D84) of cycle 1, they rolled-over to treatment cycle 2 receiving once more 3 repeated doses of AM-101 gel (0.87 mg/mL) within 5 days (D84 - D88).
- 3 Cycles AM-101: Subjects that participated in all 3 treatment cycles of the AMPACT1 study, received 3 x 3 repeated doses of AM-101 gel (0.87 mg/mL) within 5 days. The subjects could only roll-over if they completed the final follow-up of the previous cycle and were still eligible. In cycle 1 treatment was within D0 - D4. Cycle 2 treatment within D84 - D88. And treatment for cycle 3 within D168-D172. Final follow-up after 3 treatment cycles was FUV9 (D252).
Period: Overall Study
Arm/Group | 1 Cycle AM-101 | 2 Cycles AM-101 | 3 Cycles AM-101
Started | 114 | 67 | 76
Completed | 91 | 56 | 74
Not Completed | 23 | 11 | 2
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Withdrawal by Subject | 15 | 6 | 2
Not completed — Lost to Follow-up | 7 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Cycle AM-101 | 2 Cycles AM-101 | 3 Cycles AM-101 | Total
Number analyzed (Participants) | 114 | 67 | 76 | 257
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 106 | 61 | 64 | 231
  >=65 years | 8 | 6 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (14.1) | 44.7 (13.9) | 47.6 (15.5) | 44.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 17 | 21 | 63
  Male | 89 | 50 | 55 | 194
Region of Enrollment [Number; unit: participants]
  United States | 71 | 45 | 40 | 156
  Czechia | 24 | 7 | 22 | 53
  Canada | 4 | 11 | 9 | 24
  Israel | 1 | 1 | 1 | 3
  South Korea | 11 | 1 | 4 | 16
  Turkey | 3 | 2 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Subjects With a Deterioration of Hearing Threshold at Day 35 (Air Conduction)
Description: Valid for Safety Analysis Set was used.
  Air conduction: The atmospheric transmission of sound to the inner ear through the external auditory canal and via structures of the middle ear. The ability of hearing is measured in decibel (dB). The hearing threshold, is the lowest sound pressure where the ear can perceive still a sound.
  The endpoint deterioration of hearing threshold ≥15 dB in two contiguous test frequencies means that hearing worsens ≥15 dB in two neighboring sound frequencies.
Time Frame: Day 1 (TV1) to Day 35 (FUV2) of cycle 1
Population: The safety analysis set includes all subjects that had at least one intratympanic injection. Subjects are only considered at a time point if the hearing threshold is available.
Measure: Number; unit: Number subject affected
Groups:
- 1 Cycle AM-101: Subjects that participated only in 1 treatment cycle. This endpoint counts existing deteriorations at FUV2.
- 2 Cycles AM-101: Subjects that participated in 2 treatment cycles. This endpoint lists deteriorations at FUV2.
- 3 Cycles AM-101: Subjects that participated in 3 treatment cycles. This endpoint lists deteriorations at FUV2.
Arm/Group | 1 Cycle AM-101 | 2 Cycles AM-101 | 3 Cycles AM-101
Number analyzed (Participants) | 103 | 67 | 74
Number subject affected | 10 | 2 | 2
Statistical Analysis 1: Comparison: 1 Cycle AM-101 vs 2 Cycles AM-101; Fisher's exact test to assess if there is a difference in deterioration of hearing threshold between subjects that received 1 treatment cycle with AM-101 or others who received 2 treatment cycles; Test type: Superiority; p = 0.128, Fisher Exact
Statistical Analysis 2: Comparison: 1 Cycle AM-101 vs 3 Cycles AM-101; Fisher's exact test to assess if there is a difference in deterioration of hearing threshold between subjects that received 1 treatment cycle with AM-101 or others who received 3 treatment cycles; Test type: Superiority; p = 0.075, Fisher Exact
Statistical Analysis 3: Comparison: 2 Cycles AM-101 vs 3 Cycles AM-101; Fisher's exact test to assess if there is a difference in deterioration of hearing threshold between subjects that received 2 treatment cycles with AM-101 or others who received 3 treatment cycles; Test type: Superiority; p = 1, Fisher Exact

2. Primary Outcome: Frequency of Subjects With a Deterioration of Hearing Threshold at Day 119 (Air Conduction)
Description: as for outcome 1
Time Frame: Day 84 (TV4) to Day 119 (FUV5) of cycle 2
Population: The safety analysis set includes all subjects that had at least one intratympanic injection. Subjects are only considered at a time point if the hearing threshold is available.
  Subjects from Cycle 1 did not participate in Cycle 2 and 3 and are therefore "zero".
Measure: Number; unit: Number subject affected
Groups:
- 2 Cycles AM-101: Subjects that participated in 2 treatment cycles. This endpoint lists deteriorations at FUV5.
- 3 Cycles AM-101: Subjects that participated in 3 treatment cycles. This endpoint lists deteriorations at FUV5.
Arm/Group | 2 Cycles AM-101 | 3 Cycles AM-101
Number analyzed (Participants) | 59 | 75
Number subject affected | 1 | 0
Statistical Analysis 1: Comparison: 2 Cycles AM-101 vs 3 Cycles AM-101; Test type: Superiority; p = 0.4403, Fisher Exact

3. Primary Outcome: Frequency of Subjects With a Deterioration of Hearing Threshold at Day 203 (Air Conduction)
Description: as for outcome 1
Time Frame: Day 168 (TV7) up to Day 203 (FUV8) of cycle 3
Measure: Number; unit: Number subject affected
Groups:
- 3 Cycles AM-101: Subjects that participated in 3 treatment cycles. This endpoint lists deteriorations at FUV8.
Arm/Group | 3 Cycles AM-101
Number analyzed (Participants) | 74
Number subject affected | 2

4. Secondary Outcome: Frequency of Subjects With a Deterioration of Hearing Threshold at Day 84 (Air Conduction)
Description: as for outcome 1
Time Frame: Day 1 (TV1) to Day 84 (FUV3) of cycle 1
Population: as for outcome 1
Measure: Number; unit: Number subject affected
Groups:
- 1 Cycle AM-101: Subjects that participated only in 1 treatment cycle. This endpoint counts existing deteriorations at FUV3.
- 2 Cycles AM-101: Subjects that participated in 2 treatment cycles. This endpoint lists deteriorations at FUV3.
- 3 Cycles AM-101: Subjects that participated in 3 treatment cycles. This endpoint lists deteriorations at FUV3.
Arm/Group | 1 Cycle AM-101 | 2 Cycles AM-101 | 3 Cycles AM-101
Number analyzed (Participants) | 91 | 66 | 75
Number subject affected | 10 | 3 | 0
Statistical Analysis 1: Comparison: 1 Cycle AM-101 vs 2 Cycles AM-101; Test type: Superiority; p = 0.2401, Fisher Exact
Statistical Analysis 2: Comparison: 1 Cycle AM-101 vs 3 Cycles AM-101; Test type: Superiority; p = 0.0022, Fisher Exact
Statistical Analysis 3: Comparison: 2 Cycles AM-101 vs 3 Cycles AM-101; Test type: Superiority; p = 0.1001, Fisher Exact

5. Secondary Outcome: Frequency of Subjects With a Deterioration of Hearing Threshold at Day 168 (Air Conduction)
Description: as for outcome 1
Time Frame: Day 84 (TV4) to Day 168 (FUV6) of cycle 2
Population: as for outcome 1
Measure: Number; unit: Number subject affected
Groups:
- 2 Cycles AM-101: Subjects that participated in 2 treatment cycles. This endpoint lists deteriorations at FUV6.
- 3 Cycles AM-101: Subjects that participated in 3 treatment cycles. This endpoint lists deteriorations at FUV6.
Arm/Group | 2 Cycles AM-101 | 3 Cycles AM-101
Number analyzed (Participants) | 55 | 76
Number subject affected | 0 | 1
Statistical Analysis 1: Comparison: 2 Cycles AM-101 vs 3 Cycles AM-101; Test type: Superiority; p = 1.0, Fisher Exact

6. Secondary Outcome: Frequency of Subjects With a Deterioration of Hearing Threshold at Day 252 (Air Conduction)
Description: as for outcome 1
Time Frame: Day 168 (TV7) to Day 252 (FUV9) of cycle 3
Population: as for outcome 1
Measure: Number; unit: Number subject affected
Groups:
- 3 Cycles AM-101: Subjects that participated in 3 treatment cycles. This endpoint lists deteriorations at FUV9.
Arm/Group | 3 Cycles AM-101
Number analyzed (Participants) | 74
Number subject affected | 2

ADVERSE EVENTS:
Time Frame: From baseline to end of study at all visits, up to Day 252.
Description: Assessed by Investigator at all visits. In non-serious adverse events section, under occurrences (all), reported numbers are "subjects affected".
Arm/Group | 1 Cycle AM-101 | 2 Cycles AM-101 | 3 Cycles AM-101
Serious Adverse Events (participants affected / at risk) | 2/114 | 1/67 | 1/76
Other Adverse Events (participants affected / at risk) | 25/114 | 25/67 | 37/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Cycle AM-101 (N=114) | 2 Cycles AM-101 (N=67) | 3 Cycles AM-101 (N=76)
Liver function test increased (Investigations) | 1 | 0 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Cycle AM-101 (N=114) | 2 Cycles AM-101 (N=67) | 3 Cycles AM-101 (N=76)
Headache (Nervous system disorders) | 5 | 7 | 9
Ear discomfort (Ear and labyrinth disorders) | 3 | 9 | 7
Ear pain (Ear and labyrinth disorders) | 10 | 13 | 8
Hypoacusis (Ear and labyrinth disorders) | 5 | 4 | 4
Otorrhoea (Ear and labyrinth disorders) | 1 | 4 | 3
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 5
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 1
Influenza (Infections and infestations) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 4 | 2 | 6
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 | 0 | 2
Hyperacusis (Ear and labyrinth disorders) | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 1 | 2
Artificial crown procedure (Surgical and medical procedures) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees to submit a copy of any intended communication, presentation or publication (abstract, poster, article, etc.) (all together "Communication") at least 2 month in advance of the submission of proposed Communication. The Sponsor shall have 60 days, after receipt of said copies, to object to such proposed Communication. In case of such objection, the Investigator shall refrain from making such Communication for 6 months from date of receipt of such objection.